CLINICAL TRIAL: NCT00000402
Title: Long Term Effects of Calcium on Bone Mass in Young Females
Brief Title: Calcium and Bone Mass in Young Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: R01AR040736 (NIH); R01AR040736 (NIH); NIAMS-007
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Dietary calcium; Puberty; Bone density; Bone mass; Primary prevention of osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Calcium

INTERVENTIONS:
Drug: Calcium

SUMMARY:
We originally suggested that calcium in the diet is important in determining the amount of bone (bone mass) that builds up in young adults. We are testing the effect of calcium on bone mass in 354 Caucasian (white) girls. At the start of this 7-year study, the average age of the girls was 11 years, and they had not yet reached puberty. The study will also provide information about the effect of calcium on body composition (body fat) and blood pressure in young women.

We have been giving calcium to one group of participants in this study and giving a placebo (an inactive pill, or "sugar pill") to the other group. The results of this research will be important in preventing osteoporosis, because building more bone as a young person should reduce a woman's chances of developing osteoporosis later in life.

DETAILED DESCRIPTION:
This study evaluates the effect of calcium on bone mass accretion over 7 years in a cohort of 354 young females who were in pubertal Stage II at the start of the study. The average age of study participants at entry was 11 years; at the end of the study participants were 18 years old.

The study looks at skeletal development under the influence of heredity, nutrition (calcium), and physical exercise. We gave calcium to participants in one arm of this clinical trial calcium. Participants in the other arm of the trial were given a placebo. The main outcome variable is the bone mass measured at different skeletal regions.

The study will also provide data about the efficacy of calcium supplementation with regard to hypertension prevention and obesity. The results of this research will be important in preventing osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Pubertal stage II
* Calcium intake below a threshold level
* Caucasian
* Normal health

Exclusion Criteria:

* Medications affecting calcium and bone metabolism
* Chronic diseases
* Metabolic bone disease
* Abnormality in calcium metabolism

Ages: 8 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 354
Dates: Start 1991-08; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Velimir Matkovic, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- OSU Bone and Mineral Metabolism Laboratory, Columbus, Ohio, United States

REFERENCES:
- [Background] Matkovic V. Nutrition, genetics and skeletal development. J Am Coll Nutr. 1996 Dec;15(6):556-69. doi: 10.1080/07315724.1996.10718630. PMID 8951732
- [Background] Matkovic V, Ilich JZ, Andon MB, Hsieh LC, Tzagournis MA, Lagger BJ, Goel PK. Urinary calcium, sodium, and bone mass of young females. Am J Clin Nutr. 1995 Aug;62(2):417-25. doi: 10.1093/ajcn/62.2.417. PMID 7625351
- [Background] Matkovic V, Jelic T, Wardlaw GM, Ilich JZ, Goel PK, Wright JK, Andon MB, Smith KT, Heaney RP. Timing of peak bone mass in Caucasian females and its implication for the prevention of osteoporosis. Inference from a cross-sectional model. J Clin Invest. 1994 Feb;93(2):799-808. doi: 10.1172/JCI117034. PMID 8113412
- [Background] Matkovic V, Ilich JZ. Calcium requirements for growth: are current recommendations adequate? Nutr Rev. 1993 Jun;51(6):171-80. doi: 10.1111/j.1753-4887.1993.tb03097.x. PMID 8371847
- [Background] Matkovic V, Ilich J, Hsieh L. Influence of age, sex and diet on bone mass and fracture rate. Osteoporos Int. 1993;3 Suppl 1:20-2. doi: 10.1007/BF01621855. No abstract available. PMID 8461560
- [Background] Matkovic V. Calcium intake and peak bone mass. N Engl J Med. 1992 Jul 9;327(2):119-20. doi: 10.1056/NEJM199207093270210. No abstract available. PMID 1603119
- [Background] Matkovic V, Heaney RP. Calcium balance during human growth: evidence for threshold behavior. Am J Clin Nutr. 1992 May;55(5):992-6. doi: 10.1093/ajcn/55.5.992. PMID 1570810
- [Background] Matkovic V. Osteoporosis as a pediatric disease: role of calcium and heredity. J Rheumatol Suppl. 1992 Apr;33:54-9. PMID 1593603
- [Background] Matkovic V, Fontana D, Tominac C, Goel P, Chesnut CH 3rd. Factors that influence peak bone mass formation: a study of calcium balance and the inheritance of bone mass in adolescent females. Am J Clin Nutr. 1990 Nov;52(5):878-88. doi: 10.1093/ajcn/52.5.878. PMID 2239765
- [Result] Matkovic V, Landoll JD, Badenhop-Stevens NE, Ha EY, Crncevic-Orlic Z, Li B, Goel P. Nutrition influences skeletal development from childhood to adulthood: a study of hip, spine, and forearm in adolescent females. J Nutr. 2004 Mar;134(3):701S-705S. doi: 10.1093/jn/134.3.701S. PMID 14988471